CLINICAL TRIAL: NCT03642392
Title: Identification and Treatment of Early Tendinopathy in Elite Athletes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Team Denmark (Other)
Responsible Party: Principal Investigator, Christian Couppé, Senior researcher, MSc.PT, PhD., Bispebjerg Hospital
Other Study IDs: CC_1
Record Dates: First submitted 2018-08-16; First posted 2018-08-22 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Tendinopathy
Keywords: Achilles tendon; Patellar tendon; Inflammation
MeSH Terms: conditions — Tendinopathy; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tendinopathy: Athletes with unilateral tendinopathy
  Interventions: Other: Identification and treatment of early tendinopathy

INTERVENTIONS:
Other: Identification and treatment of early tendinopathy — Participants receive initial guidance about load reduction when tendinopathy

SUMMARY:
Tendon injuries represent a significant problem in elite athletes. The understanding of the pathophysiology of tendinopathy is very sparse, and especially the early events in tendinopathy are unknown. In this study, the investigators will investigate early changes in tendon tissue overloading and development of tendinopathy. The investigators will examine elite athletes with recently developed tendinopathy with regards to symptoms (pain, function), tendon morphology (ultrasonography, MRI), inflammation (the activity of inflammatory pathways) and vascularization (Doppler US). The investigators hypothesize a coupling between early symptoms and inflammatory activity, followed by structural changes. The investigation will indicate what symptoms and what tendon related measurements are primary for disease development ("tendinopathy blueprints") and should be regarding vital in the prevention of tendinopathy.

DETAILED DESCRIPTION:
The investigators intend to study the development of tendinopathy in elite athletes (badminton and handball players) that enter a phase of relative overloading of their tendons. This will be done in a large cohort of elite athletes from whom the investigators have obtained essential data and tests. A percentage of these elite athletes will develop overuse symptoms, and in those, the investigators will perform investigations that will try to identify the initial pathological changes in tendinopathy.

Participants are included as soon as possible after diagnosis of either Achilles or patellar tendinopathy because the investigators wish to investigate the early changes in tendinopathy. The hypothesis is, that at the early development of tendinopathy there will be a mismatch between matrix protein anabolic and catabolic pathways, and will be associated with a secondary upregulation of inflammatory and apoptotic markers in the tendon and result in hypervascularization and hypermetabolism.

Recruiting participants will be done in collaboration with TEAM DANMARK (the Danish sport elite sports organization) together with The Danish Badminton, Handball and Volleyball Associations). Furthermore, the investigators will establish contact with all relevant coaches and medical teams of these associations mentioned above. Information leaflets will repeatedly be sent about the project. Elite athletes can contact the chief physician of TEAM DANMARK directly through email or telephone. In comparison, a control group of healthy athletes is already recruited in the former project of recreational athletes.

Recruitment to the project will focus onset of exercise pain, and every participant will be examined by the chief physician of TEAM DANMARK if the participant has tendinopathy or not. Once included the participant will undergo following procedures as soon as possible after diagnosis is given:

* A questionnaire regarding training history and ongoing symptoms
* Ultrasound scanning of patellar or Achilles tendons (bilateral)
* Blood samples
* MRI of the tendon that can identify any diseased area.

Participants with tendinopathy will be physically reevaluated after 3, 6 and 12 months with regards to symptoms, the activity of daily life, blood samples, questionnaires VISA-A/P and ultrasound measurements. Furthermore, the unaffected side will also be used as a comparison. Moreover, participants will receive initial guidance about load reduction by the Chief Physician.

It is expected that the results of this study will provide insight into the events leading up to a developing tendinopathy. This study will add important information to understand the pathophysiology and provide information on the timing of the phases as well. Information and results from the study will give insight into better treatment options that are more specific and earlier intervention in elite athletes. Furthermore, this study will investigate and address the question of why some elite athletes develop tendinopathies, and others do not when the training volume is equally raised.

ELIGIBILITY:
Inclusion Criteria:

* Marked tendon related pain in association with exercise on one leg
* Soreness during physical examination of patellar or/and Achilles tendon upon palpation
* Demonstrate an ultrasonographic (US) thickening of the tendon on the affected side vs the contralateral un-symptomatic side in the anterior-posterior projection

Exclusion Criteria:

* • Surgery in Achilles and/or patellar tendon

  * History of Achilles and/or patellar tendinopathy
  * Received any form of an injection in Achilles and/or patella tendon
  * Lately, have an infection around Achilles and/or patella tendon

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Elite athletes 18 years and older
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2020-08-17 (Estimated); Study Completion 2021-08-17 (Estimated)

PRIMARY OUTCOMES:
Ultrasonography - Greyscale | 3 months
  Greyscale ultrasound for measuring tendon thickness (mm)
Ultrasonography - Power doppler | 3 months
  To measure tendon vascularisation, area with power doppler signal (cm^2)

SECONDARY OUTCOMES:
Measure CRP levels in blood samples 3 months follow-up | 3 months
  Systemic inflammation Whole blood, serum, plasma and tissue.
Measure CRP levels in blood samples 12 months follow-up | 12 months
  Systemic inflammation Whole blood, serum, plasma and tissue.
Tendon structural changes on MRI 3 months follow-up | 3 months
  Measure tendon structural changes on MRI
Tendon structural changes on MRI 12 months follow-up | 12 months
  Measure tendon structural changes on MRI
Ultrasonography - Greyscale | 12 months
  Greyscale ultrasound for measuring tendon thickness (mm)
Ultrasonography -Power doppler | 12 month
  To measure tendon vascularisation, area with power doppler signal (cm^2)
Victorian Institute of Sport Assessment | 3 months
  Standardised score of functional capability, in patient with achilles and patellar tendinopathy. Total score will be reported; scale (0-100). 100=full functional capacity 0=poor functional capacity.
Victorian Institute of Sport Assessment | 12 months
  Standardised score of functional capability, in patient with achilles and patellar tendinopathy. Total score will be reported; scale (0-100). 100=full functional capacity 0=poor functional capacity.
Questionnaires - Numerical Rating Scale (NRS) - Pain | 3 months
  Questions on pain, both during activity and during rest.
  Pain during activity, (NRS); Scale (0-10)
  Pain after activity, (NRS); Scale (0-10)
  Pain at rest, (NRS); Scale (0-10)
  Pain I the morning, (NRS); Scale (0-10)
  Maximal pain during the past week, (NRS); Scale (0-10)
Questionnaires - Numerical Rating Scale (NRS) - Pain | 12 months
  Questions on pain, both during activity and during rest.
  Pain during activity, (NRS); Scale (0-10)
  Pain after activity, (NRS); Scale (0-10)
  Pain at rest, (NRS); Scale (0-10)
  Pain I the morning, (NRS); Scale (0-10)
  Maximal pain during the past week, (NRS); Scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Couppé, PhD, Study Director — Unversity of Copenhagen
Locations (1):
- Institute of Sports Medicine, Copenhagen NV, Bispebjerg Hospital , København NV, Denmark

IPD SHARING:
Plan to Share IPD: No